CLINICAL TRIAL: NCT05355766
Title: Phase IIb Clinical Study to Assess the Safety and Efficacy of CN128 Tablets in the Treatment of Iron Overload in Transfusion Dependent Thalassemia With Sever Liver Iron Overloaded Patients Aged 16 and Above
Brief Title: Long-term Clinical Study of CN128 in Thalassemia With Sever Liver Iron Overloaded Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Zede Pharma-Tech Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A160605-202
Record Dates: First submitted 2022-04-22; First posted 2022-05-02 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Thalassemia; Iron Overload
MeSH Terms: conditions — Thalassemia; Iron Overload

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CN128 Group (Experimental): All subjects will be given the lower (10 mg/kg bw, bid) to higher dose (30 mg/kg bw, bid) for 52 weeks, according to the administration plan.
  The dosage form is tablets.
  Interventions: Drug: CN128 Tablets

INTERVENTIONS:
Drug: CN128 Tablets — Iron chelator, oral tablets
  Other Names: CN128

SUMMARY:
The safety and efficacy of CN128 is studied in thalassaemia with sever liver iron overloaded patients.

DETAILED DESCRIPTION:
1. The study is designed as a single arm and opened phase IIb clinical trial, so as to investigate the safety and efficacy of CN128.
2. A total of 50 eligible subjects are planned to be enrolled, and orally administration of CN128 for 52 weeks according to the administration plan.
3. Administration plan:

The trial will start with the lower dose of CN128 (10 mg/kg body weight [bw], bid) for one week. If no unacceptable toxicity associated with CN128 is found, the subjects will be given 15 mg/kg body weight [bw], bid for one week. If no unacceptable toxicity associated with CN128 is found, the subjects will be given 20 mg/kg body weight [bw], bid for two weeks. If no unacceptable toxicity associated with CN128 is found, the subjects will be given 25 mg/kg body weight [bw], bid for two weeks. If no unacceptable toxicity associated with CN128 is found, the subjects will be given 30 mg/kg body weight [bw], bid for two weeks. If no unacceptable toxicity associated with CN128 is found, the subjects will be given 30 mg/kg body weight [bw], bid to Week 52. Dosage will be adjusted according to subject status and study plan.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia patients.
* The number of blood transfusion per month ≥1. Or hemoglobin can not be maintained at 90g/L above, if blood transfusions is less than once per month.
* Severe iron overloaded patients (serum ferritin>2500 µg/L or liver iron concentration (LIC)>15 mg/g dw) despite prior treatment with at least one iron chelator.
* Patients aged 16 and above.
* Volunteer for the trial and sign the informed consent.

Exclusion Criteria:

* Active hepatitis B (HBsAg positive, HBsAb negative) or hepatitis C (HCV antibody positive, detectable HCV RNA, and Alkaline Phosphatase (ALT) beyond normal range)
* Active gastrointestinal disease history (including: gastric ulcer, duodenal ulcer, stomach or esophageal varices, ulcerative colitis, Crohn's disease, gastrointestinal cancer, familial genetic multiple intestinal polyps), and History of gastrointestinal perforation, gastrointestinal surgery that influence drug absorption, and other potential intestinal complications considered by researchers.
* ALT or Aspartate Aminotransferase (AST) > 2.5 × upper limit of normal (ULN), or serum creatinine > 1.5 × ULN.
* Neutropenia patient (neutrophil count < 1.5 × 10^9 / L).
* Active infection uncontrolled.
* Autoimmune hemolytic anemia patients.
* The patients who are currently taking CYP3A strong inducer or strong inhibitor drugs, or the drug that may extend the QT interval, or the drug that may decrease neutrophil count, but can not temporarily interrupt the use of such drugs.
* Cardiac iron overloaded patients, cardiac magnetic resonance MRI T2*<10 ms
* The patients who are allergic or contraindicated to the main ingredients or excipients of CN128 tablets.
* Congenital long QT syndrome or known family history of long QT syndrome, QTc interval>480 ms, clinically significant ventricular or atrial fast arrhythmia.
* The patients who can not accept MRI as detection means, such as claustrophobic for MRI, pacemaker, and those using ferromagnetic metal implants.
* Birth planner (including male subjects) within or within 3 months after the end of the trial.
* Participated in other clinical trials in the four weeks before taking the test preparation, except for non-interventional studies.
* Pregnant or lactating women.
* Unsuitable to participate in the trial considered by the researchers.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, adverse reactions, severe adverse events and severe adverse reactions as a measure of safety and tolerability during the study period. | Up to 52 weeks
  To determine the incidence, type and severity of adverse events, adverse reactions, severe adverse events and severe adverse reactions in patients up to 52 weeks.
Absolute Change in Weight (Unit: kg) From Baseline Over Time | Baseline, 26, 39 and 52 weeks.
  The patient's weight will be determined, and it's one kind of Physical examination.
Absolute Change in Height (Unit: m) From Baseline Over Time | Baseline, 26, 39 and 52 weeks.
  The patient's height will be determined, and it's one kind of Physical examination.
Absolute Change in Temperature (Unit: ℃）From Baseline Over Time | Baseline, 2, 4, 6, 8, 12, 16, 20, 26, 39 and 52 weeks.
  The patient's temperature will be determined, and it's one kind of vital signs checks.
Absolute Change in Blood pressure (Unit: mmHg ) From Baseline Over Time | Baseline, 2, 4, 6, 8, 12, 16, 20, 26, 39 and 52 weeks.
  Both patient's systolic and diastolic blood pressure will be measured, and it's one kind of vital signs checks.
Absolute Change in Heart rate (Unit: bpm) From Baseline Over Time | Baseline, 2, 4, 6, 8, 12, 16, 20, 26, 39 and 52 weeks.
  The patient's heart rate will be determined, and it's one kind of vital signs checks.
Absolute Change in Respiration (Unit: bpm) From Baseline Over Time | Baseline, 2, 4, 6, 8, 12, 16, 20, 26, 39 and 52 weeks.
  The patient's respiration will be determined, and it's one kind of vital signs checks.
Absolute Change in Electrocardiogram (P-R (Unit: ms), QRS (Unit: ms), QTc interval (Unit: ms), etc) From Baseline Over Time | Baseline, 2, 4, 6, 8, 12, 16, 20, 26, 39 and 52 weeks.
  The patient's electrocardiogram will be measured, and it's one kind of laboratory test.
Change in Auditory Function From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's auditory function will be determined by otorhinolaryngology.
Absolute Change in White Blood Count (Unit: 10^9/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's white blood count will be determined, and it's one kind of laboratory test.
Absolute Change in Neutrophil Count (Unit: 10^9/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's neutrophil count will be determined, and it's one kind of laboratory test.
Absolute Change in Lymphocyte Count (Unit: 10^9/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's lymphocyte count will be determined, and it's one kind of laboratory test.
Absolute Change in Monocyte Count (Unit: 10^9/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's monocyte count will be determined, and it's one kind of laboratory test.
Absolute Change in Eosinophilic Count (Unit: 10^9/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's eosinophilic count will be determined, and it's one kind of laboratory test.
Absolute Change in Basophilic Count (Unit: 10^9/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's basophilic count will be determined, and it's one kind of laboratory test.
Absolute Change in Red Blood Count (Unit: 10^9/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's red blood count will be determined, and it's one kind of laboratory test.
Absolute Change in Hemoglobin (Unit: g/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's hemoglobin will be determined, and it's one kind of laboratory test.
Absolute Change in Hematocrit (Unit:%) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's hematocrit will be determined, and it's one kind of laboratory test.
Absolute Change in Blood Platelet Count (Unit: 10^9/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's blood platelet count will be determined, and it's one kind of laboratory test.
Absolute Change in Thrombocytocrit (Unit: %) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's thrombocytocrit will be determined, and it's one kind of laboratory test.
Absolute Change in Alanine Aminotransferase (Unit: U/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's alanine aminotransferase will be determined, and it's one kind of laboratory test.
Absolute Change in Total Bilirubin (Unit:µmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's total bilirubin will be determined, and it's one kind of laboratory test.
Absolute Change in Total Protein (Unit:g/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's total protein will be determined, and it's one kind of laboratory test.
Absolute Change in Albumin (Unit: g/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's albumin will be determined, and it's one kind of laboratory test.
Absolute Change in Globulin (Unit: g/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's globulin will be determined, and it's one kind of laboratory test.
Absolute Change in Alkaline Phosphatase (Unit: U/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's alkaline phosphatase will be determined, and it's one kind of laboratory test.
Absolute Change in Aspartate Aminotransferase (Unit: U/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's aspartate aminotransferase will be determined, and it's one kind of laboratory test.
Absolute Change in Lactate Dehydrogenase (Unit: IU/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's lactate dehydrogenase will be determined, and it's one kind of laboratory test.
Absolute Change in Urea (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's urea will be determined, and it's one kind of laboratory test.
Absolute Change in Creatinine (Unit:µmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's creatinine will be determined, and it's one kind of laboratory test.
Absolute Change in Glucose (Unit: mmol/L) From Baseline Over Time [ Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's glucose will be determined, and it's one kind of laboratory test.
Absolute Change in Potassium (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's potassium will be determined, and it's one kind of laboratory test.
Absolute Change in Sodium (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's sodium will be determined, and it's one kind of laboratory test.
Absolute Change in Chlorine (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's chlorine will be determined, and it's one kind of laboratory test.
Absolute Change in Calcium (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's calcium will be determined, and it's one kind of laboratory test.
Absolute Change in Fibrinogen (Unit: g/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's fibrinogen will be determined, and it's one kind of laboratory test.
Absolute Change in Prothrombin time (Unit: s) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's prothrombin time will be determined, and it's one kind of laboratory test.
Absolute Change in Activated Partial Thromboplastin Time (APTT, Unit: s) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's APTT will be determined, and it's one kind of laboratory test.
Absolute Change in Serum Total Thyroxine (Unit: nmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's serum total thyroxine will be determined, and it's one kind of laboratory test.
Absolute Change in Parathyroid Hormone (Unit: pg/mL) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's parathyroid hormone will be determined, and it's one kind of laboratory test.
Absolute Change in Total Triiodothyronine (Unit: nmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's total triiodothyronine will be determined, and it's one kind of laboratory test.
Absolute Change in Thyrotropin (Unit: mIU/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's thyrotropin will be determined, and it's one kind of laboratory test.
Absolute Change in Urine Glucose (Unit: mmol/L) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's urine glucose will be determined, and it's one kind of laboratory test.
Absolute Change in Urine Protein (Unit: g/L)) From Baseline Over Time | Baseline, 2, 12, 26, 39 and 52 weeks.
  The patient's urine protein will be determined, and it's one kind of laboratory test.
Absolute Change in Total Testosterone (Unit: ng/ml) in men From Baseline Over Time | Baseline, 26, 39 and 52 weeks.
  The patient's total testosterone will be determined in men, and it's one kind of laboratory test.
Absolute Change in Free Testosterone (Unit: nmol/L) in men From Baseline Over Time | Baseline, 26, 39 and 52 weeks.
  The patient's free testosterone will be determined in men, and it's one kind of laboratory test.
Absolute Change in Follicle-generating Hormone (Unit: mIU/mL) in women From Baseline Over Time | Baseline, 26, 39 and 52 weeks.
  The patient's follicle-generating hormone will be determined in women, and it's one kind of laboratory test.
Absolute Change in Luteinizing Hormon (Unit: mIU/mL) in women From Baseline Over Time | Baseline, 26, 39 and 52 weeks.
  The patient's luteinizing hormonwill be determined in women, and it's one kind of laboratory test.

SECONDARY OUTCOMES:
Absolute Change in Liver iron content (Unit: mg/g dw) From Baseline Over Time | Baseline, 12, 26,39 and 52 weeks.
  Liver iron content will be determined by liver magnetic resonance.
Absolute Change in Serum ferritin (Unit: µg/L) From Baseline Over Time | Baseline, 2, 4, 6, 8, 12, 16, 20, 26, 39 and 52 weeks.
  Serum ferritin will be determined, and it's one kind of laboratory test.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Luo, PhD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital Of Guangxi Medical University, Nanning, Guangxi, China